CLINICAL TRIAL: NCT05954741
Title: Comparing the Effectiveness of Multidimensional Rehabilitation Programs for Cognitive Impairment in Comorbid Outpatients: a Randomized Controlled Trial
Brief Title: Multidimensional Rehabilitation Programs for Cognitive Impairment in Comorbid Outpatients: a Randomized Controlled Trial
Acronym: RCTCogRehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Cira Fundarò, Principal investigator, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2618 - 9.3.2022
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Impairment; Dementia; Comorbidities and Coexisting Conditions; Vascular Dementia; Dementia, Mixed
Keywords: Dementia; Comorbidity; Cognitive rehabilitation; Motor rehabilitation; Digital-based cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Dementia, Vascular; Mixed Dementias | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Patients with Neurocognitive Disorder with Clinical Dementia Rating Scale score between 0.5 and 1, due to vascular disease or due to multiple etiology), symptoms onset < 12 months, age between 65 and 80 years of age, and signed informed consent to participate in the study.
  Interventions: Other: Motor rehabilitation alone
- Group 2 (Active Comparator): Patients with Neurocognitive Disorder with Clinical Dementia Rating Scale score between 0.5 and 1, due to vascular disease or due to multiple etiology), symptoms onset < 12 months, age between 65 and 80 years of age, and signed informed consent to participate in the study.
  Interventions: Other: Motor rehabilitation and Cognitive rehabilitation (paper-based)
- Group 3 (Active Comparator): Patients with Neurocognitive Disorder with Clinical Dementia Rating Scale score between 0.5 and 1, due to vascular disease or due to multiple etiology), symptoms onset < 12 months, age between 65 and 80 years of age, and signed informed consent to participate in the study.
  Interventions: Other: Motor rehabilitation and cognitive rehabilitation (digital-based)

INTERVENTIONS:
Other: Motor rehabilitation alone — Participants will undergo motor training consisting of a walking session (20 minutes), balance exercises, postural control exercises, proprioceptive exercises, joint mobilization exercises, and muscle strengthening exercises for a total of 25 minutes. A muscle relaxation session will follow (45 minutes).
  Arms: Group 1
Other: Motor rehabilitation and Cognitive rehabilitation (paper-based) — Group 2 will perform motor training, with an analogous modality of Group 1 (45 minutes) and a standard cognitive intervention, with the execution of cognitive exercises in the domains of attention, memory, executive function, visuo-spatial abilities, space-time orientation, by paper-pencil support (45 minutes per day).
  Arms: Group 2
Other: Motor rehabilitation and cognitive rehabilitation (digital-based) — Group 3 will perform motor training, with an analogous modality of Group 1 (45 minutes) and a digital cognitive intervention, with the execution of cognitive exercises on attention, memory, executive functions, visual-spatial ability, space-time orientation, employing device support (tablet) with interactive exercises presented by specific software (VRRS Home tablet Khymeia Srl) (45 minutes).
  Arms: Group 3

SUMMARY:
Dementias secondary to cerebrovascular diseases are of significant epidemiological and clinical relevance. As a result, the management of individuals with comorbid dementia should involve early diagnosis, effective treatment, and patient-centered care planning, both in specialist and in non-specialist settings. It is well known that physical exercise can improve various aspects of health, including resistance, balance, strength, and cognitive functions such as attention and executive performance. However, the efficacy of cognitive rehabilitation is still not definitive and requires further clarification. Preliminary evidence suggests that a combination of cognitive and motor training along with novel technological approaches has the potential to maintain or improve compromised cognitive function more effectively compared to a single intervention. A multidomain intervention could enhance cognitive functioning in elderly individuals with multiple morbidities. In the present study, patients with early neurocognitive impairment based on a vascular disorder or due to multiple etiologies, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, will be screened in an outpatient multidisciplinary setting and subsequently undergo different models of rehabilitation training.

Primary aim of this study:

- Assess the effectiveness of different rehabilitation protocols for improving cognitive functions in patients with comorbid cognitive impairment. Specifically, the investigators will test the effectiveness of three rehabilitation protocols (digital-based cognitive rehabilitation combined with motor rehabilitation, paper-based cognitive rehabilitation combined with motor rehabilitation, and motor rehabilitation alone) by means of a set of multidimensional outcome measures.

Secondary aims:

- evaluating the enhancement of cognitive performance using various cognitive questionnaires categorized by cognitive domains. Additionally, the investigators will examine multidimensional variables such as motor skills, mood and anxiety levels, quality of life, patient adherence to treatment, the role of communication in patient management, caregiver burden, and the usability of digital devices (when utilized).

ELIGIBILITY:
Inclusion Criteria:

* Age Between 65 and 80 years.
* Neurocognitive Disorder due to vascular disease with Clinical Dementia Rating Scale score between 0.5 and 1, symptoms onset < 12 months.
* Neurocognitive Disorder due to multiple etiology with Clinical Dementia Rating Scale score between 0.5 and 1, symptoms onset < 12 months.

Exclusion Criteria:

* Other known neurological conditions involving cognitive functioning (e.g. Parkinson's disease, Multiple Sclerosis, head trauma, alcohol abuse).
* Severe organic instability.
* Neoplasia in progress.
* Severe psychiatric condition.
* Illiteracy.
* Severe perception deficits.
* Severe motor disability.
* Specific intellectual deficit.
* Participation in other forms of training or neurostimulation in the previous 6 months.
* Pharmacological interventions of neurological pertinence in the month before the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive performances | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  Mini Mental State Examination (Foderaro, 2022; Carpinelli Mazzi, 2020). Evaluation of various cognitive domains by answering 30 items (spatial/temporal orientation, repetition and recall of three words, working memory - backward calculation and/or spelling -, sentence repetition, sentence writing, naming, three-step command execution, constructional praxis).

SECONDARY OUTCOMES:
Changes in attention performance | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  Assessed by Trail Making Test-A, which evaluates visuospatial skills, psychomotor speed, and selective attention. In Trail Making Test A, the subject must join all 25 numbers on the sheet in ascending order in the shortest possible time.
Changes in motor performance | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  Assessed by Timed Up and Go test (TUG) (Podsiadlo & Richardson, 1991). It is a functional test to assess fall risk and static and dynamic balance. The patient is timed and asked to stand up from a chair, walk three meters, turn around, walk to the chair, and sit down. The cut-off on the total time taken in the test varies according to the clinical population observed. 6 minute walking test will be also administered ("ATS Statement: Guidelines for the Six-Minute Walk Test.," 2002). It is a simple test usually employed for assessing response to therapy in patients with pulmonary and cardiovascular disease. The test consists in walking autonomously (or held by an operator, if necessary) in a straight corridor for 6 minutes. Once the test is over, the distance traveled is calculated.
Changes in Basic Activities of Daily Living | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Basic Activity of Daily Living (BADL) (Katz et al., 1963) is a scale for assessing basic activities related to everyday living. The scale proposes 6 basic activities (bathing; dressing; toileting; continence; moving; feeding). At the end of the assignment, the total score is calculated by summing all the points from each item.
Changes in Instrumental Activities of Daily Living | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Instrumental Activity of Daily Living (IADL) (Lawton & Brody, 1969). It is used to assess the levels of autonomy in life activities (basic and instrumental) of the patient by the caregiver. Thus, 8 complex functions are reported (using the telephone; shopping; using transportation; cooking (women only); doing housework (women only); doing laundry (women only); handling money; taking medications).
Changes in Anxious Symptoms | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Generalized Anxiety Disorder-7 (GAD) (Spitzer et al., 2006) is a questionnaire built to measure the severity of anxiety symptoms in the previous two weeks.
Changes in Depressive Symptoms | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Patient Health Questionnaire-9 (PHQ-9) (Spitzer et al., 1999) is a scale currently used in general practice to determine the diagnosis, severity, and subsequent monitoring of depressive conditions in patients.
Changes in Neuropsychiatric Symptoms | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Neuropsychiatric Inventory NPI-Q (Kaufer et al., 2000) is a self-report questionnaire administered to the caregiver in order to assess the occurrence and severity of a range of neuropsychiatric symptoms in the patient during the past few weeks.
Changes in Caregiver Burden | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Family Strain Questionnaire (FSQ) - Short Form (FSQ-SF) (Ferrario et al., 2004) is a screening tool that aims to gather information on the situation experienced by a primary caregiver in the care setting, such as emotional overload, and organizes its scores according to areas of increasing criticality.
Changes in Health-Related Quality of Life (Questionnaire) | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The EuroQol 5D-5L (Rabin & de Charro, 2009). It is a questionnaire consisting of 5 sections (motor abilities; personal care; usual activities; pain; anxiety and depression) and provides the option to select a level of severity (1, no problem; 2, moderate problem; 3, severe problem).
Changes in Health-Related Quality of Life (Visual Analogue Scale) | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The EuroQol 5D-5L - VAS (Rabin & de Charro, 2009). The EuroQoL Visual Analogue Scale (EQ VAS) consists of a visual analogue scale from 0 (Worst imaginable health state) to 100 (Best imaginable health state), where the subject is asked to indicate the level of self-perceived wellness.
Changes in Treatment Adherence | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Morisky Green Levine (MGL) Adherence Scale (Morisky et al., 1986) is a rapidly administered questionnaire widely used to assess nonadherence to medication prescriptions. Its 4-item version consists of 4 questions with strictly behavioral content that can be answered in binary form (yes/no). The content of the questions varies from forgetfulness and inattention in taking the medication to autonomous discontinuation of the prescription without the doctor's permission.
Changes in HealthCare Communication | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  The Communication Assessment Tool (CAT) (Scala et al., 2016) is a 15-item questionnaire created to assess patients' perceptions of the physician's communication effectiveness. Patients are asked to respond based on a single encounter with the physician.
Changes in System Usability (for Group 3 exclusively) | Evaluation performed at baseline (pre-intervention), post-intervention (after 8 weeks) and at follow up (after 3 months).
  Changes in System Usability will be addressed with the SUS scale. The System Usability Scale (SUS) (Kortum et al., 2020) consists in a self-reported assessment of the degree of perceived usability as a result of using a wide variety of devices and systems. The higher the scores, the higher the degree of perceived usability. The score ranges from A=excellent usability to F=poor usability based on the normal distribution of the percentile range of mean scores: A = >80.3; B = 80.3-68; C = 68; D = 67-51; F = <51.
  It consists of 10 items on a 5-point Likert scale (1=not at all agree; 5=fully agree). The range for scoring each item is 0-4. The total scores are between 0 and 100 and are obtained by subtracting the raw scores at items 1, 3, 5, 7, and 9 by one, while the raw scores at items 2, 4, 6, 8, and 10 will be subtracted from 5. The adjusted scores are added together and the total sum is multiplied by 2.5, thus obtaining the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri - Montescano, Montescano, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fundaro C, Granata N, Traversoni S, Torlaschi V, Maestri R, Maffoni M, Baiardi P, Grossi F, Buonocore M, Gabanelli P, Manera MR, Pierobon A. Multidimensional screening and intervention program for neurocognitive disorder in vascular and multimorbid outpatients: Study protocol for a randomized clinical trial. PLoS One. 2024 Jul 10;19(7):e0306256. doi: 10.1371/journal.pone.0306256. eCollection 2024. PMID 38985746